CLINICAL TRIAL: NCT07406776
Title: Identification of Histories of Pregnancy Termination, Particularly Early Miscarriage, in General Medical Records.
Status: Completed | Type: Observational
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2024_RIPH_07_DMG-Fausse couche
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Early Miscarriage
Keywords: early miscarriage; termination pregnancy; general medical
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early miscarriage (EM) is defined as the spontaneous expulsion of an intrauterine pregnancy of less than 14 weeks' duration. Early miscarriage is a very common complication, affecting more than 10% of pregnancies. Because of its frequency, EM is often considered a trivial event, particularly by healthcare professionals.

However, for the women who experience it, EM can be a traumatic event, difficult to discuss with their families, and a source of worries and questions for subsequent pregnancies. The international literature is consistent on the psychological morbidity associated with miscarriage: anxiety, depression and post-traumatic stress disorder have been studied in women following CPT. The identification of a history of EM by doctors is therefore important for the overall management of women's health.

The 2021 National Perinatal Survey showed that less than 5% of pregnant women in France had their first six months of pregnancy monitored by a general practitioner, a proportion that has been steadily declining in recent years. The majority of women are monitored by a gynecologist, or in 40% of cases by a midwife. These professionals therefore appear to be the preferred point of contact for women in the event of a miscarriage. In the absence of specific information, either from the woman herself or from the healthcare professional who treated her, the general practitioner-the attending physician may remain unaware of this event in their patient's life. Under these circumstances, identifying a history of EM in the general practitioner's medical records may not be sufficient.

DETAILED DESCRIPTION:
The primary objective is to describe the frequency of notification of a history of early miscarriage in the treating physician's medical record.

The secondary objectives are :

* To describe how the treating physician is informed of the history of early miscarriage.
* To investigate the factors associated with notification of a history of early miscarriage in the treating physician's medical record medical records.
* Describe the frequency of notification of a history of termination of pregnancy other than early miscarriage (voluntary termination of pregnancy, foetal death in utero, medical termination of pregnancy) in the treating physician's medical record.
* Describe the procedures for informing the attending doctor about the history of termination of pregnancy other than early miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged between 18 and 50
* Whose GP has agreed to take part in the study
* Agreeing to take part in the study.

Exclusion Criteria:

* Minors
* Over the age of 50
* Protected by law (guardianship, curatorship, safeguard of justice)
* Refusing to take part in the study.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Women aged between 18 and 50, who declared a GP participating in the study as their GP and agreed to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2026-02-05 (Actual)

PRIMARY OUTCOMES:
notification of early miscarriage in the medical file of the woman who reported it. | Day 0
  the frequency of notification of a history of early miscarriage in the attending physician's medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Gestonnairedu CURRS, Reims, Champagne-Ardenne, France